CLINICAL TRIAL: NCT00407459
Title: Phase II Study of the Combination of Bevacizumab Plus Pemetrexed and Carboplatin as First-line Therapy in Patients With Malignant Pleural Mesothelioma
Brief Title: Phase II Study of Bevacizumab, Pemetrexed and Carboplatin as First-Line Therapy in Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Armando Santoro, MD (Other)
Responsible Party: Sponsor-Investigator, Armando Santoro, MD, MD, Istituto Clinico Humanitas
Organization: Istituto Clinico Humanitas (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2006-003; EUDRACT 2006-004429-27
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — Bevacizumab; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Bevacizumab, Pemetrexed, Carboplatin — * Bevacizumab: 15 mg/kg intravenous infusion over 30 to 90 minutes, following chemotherapy, on Day 1 every 3 weeks
  * Pemetrexed: 500 mg/m2 intravenous infusion over 10 minutes on Day 1 every 3 weeks
  * Carboplatin: AUC 5 intravenous infusion over 1 hour on Day 1 every 3 weeks
  Other Names: Avastin; Alimta; Carboplatin

SUMMARY:
The primary objective is to assess antitumor activity of the combination of bevacizumab, pemetrexed and carboplatin, in terms of time to progression.

DETAILED DESCRIPTION:
Secondary endpoints are to evaluate:

* the objective response rate (RR) of the combination;
* the toxicity and the safety profile of the combination;
* the duration of response (RD) and time to treatment failure (TTF);
* the overall survival (OS)
* RR, TTP and OS according to baseline plasma VEGF levels (introduced with Amendment 1 dated 8/11/2007)

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven malignant pleural mesothelioma, inoperable, non previously treated with chemotherapy including intracavitary administration
* PS 0-1
* Measurable and/or evaluable lesions according to RECIST criteria
* Adequate organ function

Exclusion Criteria:

* Uncontrolled hypertension
* Evidence of bleeding diathesis or coagulopathy
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2007-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Time to progression (TTP) from first day of treatment until first observation of disease progression or death due to any cause or the last date the patient was known to be progression free or alive. | At the end of study

SECONDARY OUTCOMES:
Response rate (RR) assessed according to modified RECIST criteria for Malignant Pleural Mesothelioma. | Two months after the end of enrollment
Overall survival (OS) computed as the time between the first day of treatment and the date of death or the last date the patient was known to be alive. | At the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy

REFERENCES:
- [Background] Ceresoli GL, Zucali PA, Favaretto AG, Grossi F, Bidoli P, Del Conte G, Ceribelli A, Bearz A, Morenghi E, Cavina R, Marangolo M, Parra HJ, Santoro A. Phase II study of pemetrexed plus carboplatin in malignant pleural mesothelioma. J Clin Oncol. 2006 Mar 20;24(9):1443-8. doi: 10.1200/JCO.2005.04.3190. PMID 16549838
- [Background] Ceresoli GL, Chiti A, Zucali PA, Rodari M, Lutman RF, Salamina S, Incarbone M, Alloisio M, Santoro A. Early response evaluation in malignant pleural mesothelioma by positron emission tomography with [18F]fluorodeoxyglucose. J Clin Oncol. 2006 Oct 1;24(28):4587-93. doi: 10.1200/JCO.2006.06.8999. PMID 17008700
- [Derived] Ceresoli GL, Zucali PA, Mencoboni M, Botta M, Grossi F, Cortinovis D, Zilembo N, Ripa C, Tiseo M, Favaretto AG, Soto-Parra H, De Vincenzo F, Bruzzone A, Lorenzi E, Gianoncelli L, Ercoli B, Giordano L, Santoro A. Phase II study of pemetrexed and carboplatin plus bevacizumab as first-line therapy in malignant pleural mesothelioma. Br J Cancer. 2013 Aug 6;109(3):552-8. doi: 10.1038/bjc.2013.368. Epub 2013 Jul 16. PMID 23860535